CLINICAL TRIAL: NCT03636737
Title: Retrospective Multicenter Observational Study on the Clinical Features, Comorbidities and Pathologies Associated With Pyoderma Gangrenosum in Patients Diagnosed With This Pathology Between 2000 and 2015
Brief Title: Study on the Clinical Features, Comorbidities and Pathologies Associated With Pyoderma Gangrenosum
Acronym: PYODERMA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: RCAPHM17_0083
Record Dates: First submitted 2018-08-16; First posted 2018-08-17 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Pyoderma Gangrenosum
MeSH Terms: conditions — Pyoderma Gangrenosum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- experimental group: Patients with Pyoderma gangrenosum
  Interventions: Other: pathology associated

INTERVENTIONS:
Other: pathology associated — list of pathology associated to Pyoderma gangrenosum

SUMMARY:
Pyoderma gangrenosum (PG) is a rare disease. She is often under diagnosed and a source of diagnostic wandering and inadequate care. Moreover, its association in more than one case out of two to a significant underlying pathology, such as inflammatory bowel disease, inflammatory rheumatism, or hematology, makes its diagnosis essential. Its pathophysiological mechanisms remain controversial and many other comorbidities have been reported in the literature, including endocrinological, cardiovascular and metabolic, neoplastic and autoimmune comorbidities.

The objective is to study the field, comorbidities and pathologies associated with PG on a series of patients diagnosed with PG, as well as to characterize the clinical and histological aspects of lesions.

A retrospective observational non-interventional multicenter study is proposed. 10 French centers. The recruitment will be done via the DIM using coding software: codes L984 , L982 and L97 according to 2 major criteria (typical clinical appearance with ulceration well limited and purulent or pustule hutches, exclusion of differential diagnoses) and at least 2 minor criteria (among compatible histological aspect, classically compatible associated pathologies, corticosensitivity of lesions, pathergie phenomenon, painful lesions).

Demographic data, clinical appearance of the lesions, cardiovascular and metabolic comorbidities, other associated pathologies, histological findings of the ulcer biopsy and biological results to describe the population and associated pathologies or comorbidities to PG

DETAILED DESCRIPTION:
Pyoderma gangrenosum (PG) is a rare disease. She is often under diagnosed and a source of diagnostic wandering and inadequate care. Moreover, its association in more than one case out of two to a significant underlying pathology, such as inflammatory bowel disease, inflammatory rheumatism, or hematology, makes its diagnosis essential. Its pathophysiological mechanisms remain controversial and many other comorbidities have been reported in the literature, including endocrinological, cardiovascular and metabolic, neoplastic and autoimmune comorbidities.

The objective is to study the field, comorbidities and pathologies associated with PG on a series of patients diagnosed with PG, as well as to characterize the clinical and histological aspects of lesions.

A retrospective observational non-interventional multicenter study is proposed. 10 French centers. The recruitment will be done via the DIM using coding software: codes L984 (chronic skin ulceration), L982 (febrile neutrophilic dermatosis) and L97 (leg ulcer) according to 2 major criteria (typical clinical appearance with ulceration well limited and purulent or pustule hutches, exclusion of differential diagnoses) and at least 2 minor criteria (among compatible histological aspect, classically compatible associated pathologies, corticosensitivity of lesions, pathergie phenomenon, painful lesions).

Demographic data, clinical appearance of the lesions, cardiovascular and metabolic comorbidities, other associated pathologies, histological findings of the ulcer biopsy and biological results to describe the population and associated pathologies or comorbidities to PG

ELIGIBILITY:
Inclusion Criteria:

* 2 major criteria (typical clinical appearance with well-defined ulceration and purulent or pustule hutches, exclusion of differential diagnoses)
* at least 2 minor criteria (among compatible histological aspect, classically compatible associated pathologies, corticosensitivity of the lesions, pathergie phenomenon, painful lesions).

Exclusion Criteria:

* patients with less than 2 major criteria
* patients with less than 2 minor criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with pyoderma gangrenosum
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients | 1 months
  Number of patients with Pyoderma gangrenosum and associated pathology

CONTACTS AND LOCATIONS:
Overall Officials: EMILIE GARRIDO PRADALIE, Study Director — APHM
Locations (1):
- Assistance Publique Des Hopitaux de Marseille, Marseille, PACA, France